CLINICAL TRIAL: NCT00202527
Title: Efficacy of the Treatment With Nasal Positive Continuous Airway Pressure to Reduce the Arterial Blood Pressure in Patients With Apneas-Hypopneas During the Sleep and Systemic Hypertension
Brief Title: Spanish Cohort for the Study of the Effect of CPAP in Hypertension (CEPECTA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI041110
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-12-23 (Estimated); Status verified 2005-09

CONDITIONS: Sleep Apnea; Hypertension
Keywords: Sleep apnea; Hypertension; CPAP
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypertension

INTERVENTIONS:
Device: Nasal continuos positive airway pressure

SUMMARY:
AIMS:To know the effects of the treatment with nasal positive continuous airway pressure (CPAP) on systemic blood pressure and the expression of biological mediators, in systemic hypertension of recent diagnostic, whose have an apnea-hypopnea index > 15.

METHODOLOGY: DESIGN: Prospective, multicenter, randomized study, of parallel groups and controlled with placebo, in patients diagnosed of systemic hypertension (SH) with an apnea-hypopnea index, by conventional polysomnography > 15. A total of 340 patients with recently diagnosed of SH and without any pharmacological treatment will be studied. All patients will be randomized to receive, alternatively, CPAP treatment with optimal pressure titled with a proved system, or Sham-CPAP for 12 weeks.

MEASUREMENTS: A) Conventional polysomnography at baseline: B) Clinic: sleepiness (ATS, Basic Nordic Sleep Questionnaire and Epworth), quality of life (EuroQol); C) 24 hour blood pressure monitoring; D) Expression of biological mediators in blood: general determinations, endothelial, inflammatory, lipid, renin-angiotensin-aldosterone and adrenergic mediators.

ANALYSIS. Baseline measurements of all the variables will be compared with the situation at six and twelve weeks. We will use the chi square test and the Fisher´s exact test (categorical variables), the t test for continous variables and repeated measures ANCOVA for the primary objective. The analyses will be done under the criterion of intention to treat and for protocol. The variables will be controlled by the compliance with the CPAP..

ELIGIBILITY:
Inclusion Criteria:

* Patients, both sexes from 18 to 75 years old, with clinical suspected of OSAH defined by an apnea-hypopnea index > 15 and having a recent diagnosis of hypertension which have not received any pharmacological treatment for hypertension.

Exclusion Criteria:

Inclusion Criteria:

* Patients with clinical suspected of OSAH defined by an apnea-hypopnea index > 15 and having a recent diagnosis of hypertension which have not received any pharmacological treatment for hypertension.

Exclusion Criteria:

* Severe excessive daytime sleepiness; professional drivers; pregnant women; alcohol consumption more than 100 gr. Ethanol per day; sedative medication; psychiatric illness; malignant or complicated hypertension; renal insufficiency; severe chronically ilness or malignant ilness; severe craniomandibular disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340
Dates: Start 2005-01; Study Completion 2005-09

PRIMARY OUTCOMES:
Effect of CPAP in 24 hours blood pressure monitoring
effect of CPAP y quality of life and clinical aspects

SECONDARY OUTCOMES:
effect of CPAP in biologic mediators

CONTACTS AND LOCATIONS:
Overall Officials: JOAQUIN DURAN-CANTOLLA, MD, Principal Investigator — Sociedad Española de Cirugía Torácica
Locations (1):
- Unit of Research. Hospital Txagorritxu, Vitoria-Gasteiz, ALAVA, Spain

REFERENCES:
- [Derived] Duran-Cantolla J, Aizpuru F, Montserrat JM, Ballester E, Teran-Santos J, Aguirregomoscorta JI, Gonzalez M, Lloberes P, Masa JF, De La Pena M, Carrizo S, Mayos M, Barbe F; Spanish Sleep and Breathing Group. Continuous positive airway pressure as treatment for systemic hypertension in people with obstructive sleep apnoea: randomised controlled trial. BMJ. 2010 Nov 24;341:c5991. doi: 10.1136/bmj.c5991. PMID 21106625